CLINICAL TRIAL: NCT06042946
Title: Microsurgical Resection of Intramedullary Spinal Cord Metastases - a Retrospective International Multicenter Study
Brief Title: Microsurgical Resection of Intramedullary Spinal Cord Metastases
Status: Recruiting | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: University Hospital, Zürich (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Geneva (Other); Kantonsspital Aarau (Other); Kantonsspital Winterthur KSW (Other); Luzerner Kantonsspital (Other); Klinikum rechts der Isar Technische Universität München (Unknown); University Hospital Muenster (Other); University of Toronto (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Felix C. Stengel, MD, Junior Attending Neurosurgeon, Cantonal Hospital of St. Gallen
Other Study IDs: 2023-00292
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Metastasis; Spinal Cord Tumor Malignant Intramedullary; Functional Outcome; Radiotherapy; Complications; Spinal Cord Neoplasms
Keywords: Spinal cord metastasis
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- iscm_resection: -Adult patients admitted to one of the participating centres and treated for ISCM between 2017 and 2023 by resection of the ISCM with or without adjuvant radiotherapy
  Interventions: Procedure: Microsurgical resection of ISCM
- iscm_radiotherapy: -Adult patients admitted to one of the participating centres and treated for ISCM between 2017 and 2023 by radiotherapy without resection of the ISCM

INTERVENTIONS:
Procedure: Microsurgical resection of ISCM — Microsurgical resection of ISCM defines the surgical removal of cancerous tumors that have spread to the spinal cord, using advanced microsurgical techniques and equipment like ultrasound, neuromonitoring, ultrasonic aspirator to prevent damage to the spinal cord.
  Groups: iscm_resection

SUMMARY:
The aim of the study is to establish a multi-center, retrospective database for patients with intramedullary spinal cord metastases (ISCM) and analyse the functional outcome in surgically treated ISCM patients.

The hypothesis is that the surgical treatment of selected ISCM patients does not lead to persistent morbidity and does not increase mortality, compared to patients that are treated non-operatively.

Secondary objectives are to assess pre- to postoperative neurological deficits, ambulatory status, and overall survival of surgically treated ISCM patients.

The investigators intend to include a control cohort of patients with ISCM from participating centers, who underwent non-surgical oncological treatment (radiotherapy with or without chemotherapy). This control cohort of patients will be used to match patients with and without surgical treatment.

Primary endpoint (analysed in surgically treated ISCM patients):

Functional outcome at 90 days after treatment initiation, measured by the modified McCormick Scale. This is a score for grading of neurological function in spinal cord conditions.

The McCormick scale ranges from Grade I (neurologically intact) to grade V (paraplegic or quadriplegic). The McCormick scale is suitable for our retrospective study because of its good reproducibility and comparability.

Secondary endpoints (analysed in surgically treated ISCM patients and analysed in matched patients with and without surgical treatment):

* Functional outcome by the McCormick scale and the modified Japanese Orthopaedic Association scale (mJOA) at 6 and 12 months. This is a score evaluating motor function of upper and lower extremities, sensory function of upper extremities and sphincter function / voidance. The mJOA ranges from 0 - 18 points, with higher score values representing better functional outcome. The minimum clinically important difference of the mJOA is 1-2 points, and scores lower than 14 indicate moderate myelopathy, scores lower than 11 indicate severe myelopathy.
* Ambulatory status and continence at 90 days, 6 & 12 months (determined by mJOA subscores)
* Neurological outcome, measured by American Spinal Cord Injury Association (ASIA)
* Impairment Scale at 90 days, 6 and 12 months
* Rate & type of complications at 90 days after treatment according to The Novel Therapy
* Disability-Neurology Grade (TDN grade)16
* Overall survival (in days)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to one of the participating centres and treated for ISCM
* Available documentation of admission and postoperative status

Exclusion Criteria:

- Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who have undergone treatment for ISCM at one of the participating hospitals in the period from 2017 to 2023. The study period is chosen, as electronic documentation is available at all hospitals in this time-period. Patients will be identified by generated lists from neurosurgery (microsurgical procedures for ISCM) and radiooncology (radiotherapy for ISCM).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome at 90 days after treatment initiation | at 90 days after treatment initiation
  measured by the modified McCormick Scale. This is a score for grading of neurological function in spinal cord conditions.
  The McCormick scale ranges from Grade I (neurologically intact) to grade V (paraplegic or quadriplegic). The McCormick scale is suitable for our retrospective study because of its good reproducibility and comparability.

SECONDARY OUTCOMES:
Functional outcome | at 3, 6 and 12 months after treatment initiation
  modified Japanese Orthopaedic Association Score (mJOA) Range 0-18, with lower scores indicate a more sever myelopathy
Neurological outcome | at 6 and 12 months after treatment initiation
  measured by American Spinal Cord Injury Association (ASIA) Impairment Scale (AIS) A: Complete. No sensory or motor function is preserved in sacral segments S4-S5, no sacral sparing B: Sensory Incomplete. Sensory but not motor function is preserved below the neurological level and includes sacral segments S4-S5, AND No motor function is preserved more than three levels below the motor level on either side of the body C: Motor Incomplete. Motor function is preserved below the neurological level AND More than half of the key muscle functions below the neurological level of injury have a muscle grade of less than 3 (Grades 0-2) D: Motor Incomplete. Motor function is preserved below the neurological level AND At least half (half or more) of the key muscle functions below the neurological level of injury have a muscle grade ≥ 3 E: Normal. If sensation and motor function are graded as normal in all segments AND the patient had prior SCI-related deficits
Rate & type of complications | within 90 days after treatment initiation
  Therapy-Disability-Neurology Grade (TDN Grade) Range: Grade 1-5 The Therapy-Disability-Neurology (TDN) grading system is a novel multidimensional classification of complications severity.
  higher Grades indicate higher severity of complication
Functional outcome | at 6 and 12 months after treatment initiation
  measured by the modified McCormick Scale. This is a score for grading of neurological function in spinal cord conditions.
  The McCormick scale ranges from Grade I (neurologically intact) to grade V (paraplegic or quadriplegic). The McCormick scale is suitable for our retrospective study because of its good reproducibility and comparability.

CONTACTS AND LOCATIONS:
Overall Officials: Martin N. Stienen, PD, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St. Gallen, Neurosurgery, Sankt Gallen, Switzerland